CLINICAL TRIAL: NCT04342143
Title: Reliability and Validity of the Vicorder Device When Measuring Pulse Wave Velocity and Transit Time Within Chronic Stroke Patients
Brief Title: Reliability and Validity of the Vicorder Device When Measuring Pulse Wave Velocity Within Chronic Stroke Patients
Status: Recruiting | Type: Observational
Sponsor: University of Winchester (Other)
Responsible Party: Sponsor
Other Study IDs: Paine_Validity_VIC
Record Dates: First submitted 2020-04-08; First posted 2020-04-10 (Actual); Last update posted 2024-05-17 (Actual); Status verified 2024-05

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke | interventions — Blood Pressure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

GROUPS / COHORTS (1):
- Stroke: Patients who have a diagnosis of stroke by a stroke consultant from UK National Health Service Trust within 3 months to 5 years of study start date.
  Interventions: Device: Blood pressure and ultrasound assessment

INTERVENTIONS:
Device: Blood pressure and ultrasound assessment — No intervention. Participants will undertake an overnight fast prior to each assessment (only water is allowed to be consumed prior to the assessment). Participants will be asked to visit the lab on four separate occasions; the first two sessions will involve triplicated measures of carotid-femoral PWV (cfPWV), brachial-femoral PWV (bfPWV), brachial-ankle PWV (baPWV), femoral-ankle PWV (faPWV) and TT by the Vicorder in both seated and supine position. The SphygmoCor will also be used to assess cfPWV in both seated and supine. During the third and fourth sessions individuals will be randomised into either a supine or seated position. A 3 lead ECG will be attached and ultrasound video clips will be taken at the carotid, brachial, femoral and posterior tibial artery on both the symptomatic and asymptomatic sides to look at stiffness and blood velocity. Following this, the Vicorder will be used to look at cfPWV, bfPWV, baPWV, faPWV and TT on both sides.

SUMMARY:
Stroke is a major global health problem and main cause of disability worldwide. Blood pressure control is important for good health in stroke patients. Measuring central blood pressure (the blood pressure which is found in the heart) and measuring the stiffness of your arteries will give practitioners, clinicians and researcher's important information over and above what is usually obtained from peripheral blood pressure in the arm. The most validated and most recognisable equipment for central blood pressure and arterial stiffness is the SphygmoCor XCEL. However, the Doppler Ultrasound is used more often in population-based studies and has been shown to be a precise and accurate measurement. Although these devices are validated, they both require a highly skilled operator and are quite time-consuming. As such, it is important to explore less operator dependent and time consuming devices, such as the Vicorder, as this could be essential for researchers and clinicians.Therefore, this study will investigate whether the Vicorder device is valid and reliable when measuring these outcomes and if so could be implemented in large research studies and potenially be used by clinicians.

DETAILED DESCRIPTION:
Twenty stroke patients will be recruited for this study. Participants will take part in four seperate assessments (2 hours each) with a minimum of 24 hour recovery between each session. Before each assessment participants will undertake an overnight fast (only water is allowed to be consumed prior to the assessment). If required, participants will take their medication the morning of each assessment and this will be noted.During the first session participants will be randomised into either a supine or seated condition. Participants will rest in this posture for 15 minutes. Triplicate measures of peripheral blood pressure and pulse wave analysis will be measured using the SphygmoCor XCEL and Vicorder device. A 3-lead ECG will be placed on the participant and ultrasound measures will be taken at the carotid, brachial, femoral and posterior tibial artery. This will examine the caroid-femoral pulse wave velocity (cfPWV), brachial-femoral pulse wave velocity (bfPWV), brachial-ankle pulse wave velocity (baPWV) and femoral-ankle pulse wave velocity (faPWV). Following this, the Vicorder device will be used to measure these segments. All measures will be on both symptomatic and asymptomatic sides. This procedure will be repeated in a seperate session whereby individuals will be in the other posture.

Session 3 and 4 will include participants resting for 15 minutes in a supine position. Triplicate measures of peripheral blood pressure and pulse wave analysis will be taken with the Vicorder. Followed by triplicate measures of cfPWV, bfPWV, baPWV and faPWV. This will be repeated in a seated position within the same session.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of stroke by a stroke cnsultant from a UK National Health Service Foundation Trust
* 3 months to 5 years of study start date

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients diagnosed with stroke by a stroke consultant at a local hospital will be eligible to participate.
Sampling Method: Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2020-03-01 (Actual); Primary Completion 2024-06 (Estimated); Study Completion 2024-06 (Estimated)

PRIMARY OUTCOMES:
Pulse Wave Velocity | 1 month
  Pulse wave velocity will be assessed on four seperate days in both seated and supine posture. This will be measured with the Vicorder, Ultrasound & SphygmoCor
Transit Time | 1 month
  Transit time will be assessed on four seperate days in both seated and supine posture. This will be measured with the Vicorder, Ultrasound & SphygmoCor

SECONDARY OUTCOMES:
Peripheral blood pressure | 1 month
  Peripheral blood pressure will be measured on four seperate days in both supine and seated posture. This will be meausred with the SphygmoCor and Vicorder.
Pulse wave analysis | 1 month
  Pulse wave analysis will be measured on four seperate days in both supine and seated posture. This will be meausred with the SphygmoCor and Vicorder.

CONTACTS AND LOCATIONS:
Locations (1):
- Physiology Laboratory, Winchester, United Kingdom

IPD SHARING:
Plan to Share IPD: No